CLINICAL TRIAL: NCT04150887
Title: An Open-label, Multicenter, Phase 1b Study of OV-1001 (Cusatuzumab; Anti-CD70 Monoclonal Antibody) in Combination With Background Therapy for the Treatment of Subjects With Acute Myeloid Leukemia
Brief Title: Cusatuzumab in Combination With Background Therapy for the Treatment of Participants With Acute Myeloid Leukemia
Acronym: ELEVATE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OncoVerity, Inc. (Industry)
Collaborators: argenx (Industry); Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELEV20235; 2019-002808-41 (EudraCT Number); ELEV20235 (Other: OncoVerity, Inc.); 74494550AML1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Cohort 2: Cusatuzumab + Venetoclax (Experimental): Participants enrolled in this cohort will receive venetoclax ramp-up to 400 mg orally (as background therapy) starting on Cycle 1 Day 1 and followed by 400 mg daily dosing starting on Cycle 1 Day 4 plus cusatuzumab IV on Day 3 and Day 17 of each 28-day cycle. Cohort 2 will not be enrolled in the US.
  Interventions: Drug: Cusatuzumab; Drug: Venetoclax
- Cohort 3: Cusatuzumab + Venetoclax + Azacitidine (CVA) (Experimental): Participants enrolled at US sites will receive cusatuzumab 10 mg/kg and potentially escalate to 20 mg/kg IV in combination with azacitidine 75 mg/m^2 SC or IV plus venetoclax ramp-up to 400 mg orally (as background therapies). Participants enrolled from ex-US sites will receive cusatuzumab 20 mg/kg and potentially de-escalate to 10 mg/kg IV in combination with azacitidine 75 mg/m^2 SC or IV plus venetoclax ramp-up to 400 mg orally (as background therapies).
  Interventions: Drug: Cusatuzumab; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Cusatuzumab — Cusatuzumab will be administered as a dose of 10mg/kg or 20mg/kg intravenously.
  Other Names: JNJ-74494550; ARGX-110
Drug: Azacitidine — Azacitidine will be administered 75 mg/m^2 subcutaneously or intravenously.
  Other Names: Vidaza
  Arms: Cohort 3: Cusatuzumab + Venetoclax + Azacitidine (CVA)
Drug: Venetoclax — Venetoclax will be administered orally and the dose will ramp-up to 400 mg.
  Other Names: Venclexta

SUMMARY:
The purpose of the study is to characterize safety and tolerability of cusatuzumab in combination with various therapies used to treat acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) according to World Health Organization 2016 criteria . Participants with acute promyelocytic leukemia (APL) are not eligible
* Must be ineligible for intensive chemotherapy
* De novo or secondary AML
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Previously untreated AML except: emergency leukapheresis, hydroxyurea, and/or 1 dose 1-2 gram per meter square (g/m^2) cytarabine during the Screening Phase to control hyperleukocytosis. These treatments must be discontinued greater than or equal to (>=) 24 hours prior to start of study drug. Empiric all trans retinoic acid (ATRA) treatment for presumed acute promyelocytic leukemia (APL) is permitted but APL must be ruled out and ATRA must be discontinued >=24 hours prior to the start of study drug
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies

Exclusion Criteria:

* Leukemic involvement of the central nervous system
* Eligible for an allogeneic hematopoietic stem cell transplantation at study entry
* Received a live, attenuated vaccine within 4 weeks prior to initiation of study drug
* A history of human immunodeficiency virus (HIV) antibody positive or tests positive for HIV if tested at screening
* Known allergies, hypersensitivity, or intolerance to cusatuzumab, venetoclax, azacitidine, or their excipients (example: mannitol, an excipient of azacitidine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Frequency and Severity of Adverse Events (AEs), Laboratory Abnormalities, and Physical Exam Findings as a Measure of Safety | Up to 42 months
  Frequency and severity of AEs, laboratory abnormalities, and physical exam findings will be reported.

SECONDARY OUTCOMES:
Serum Concentration of Cusatuzumab | Up to 23 months
  Serum concentration of cusatuzumab will be assessed.
Number of Participants with Anti-cusatuzumab Antibodies | Up to 23 months
  Number of participants with anti-drug antibodies to cusatuzumab will be reported.
Percentage of Participants with Complete Response (CR) | Up to 42 months
  Percentage of participants with complete response based on European Leukemia Network (ELN) 2017 response criteria assessment will be reported.
Percentage of Participants with Complete Remission with Partial Hematological Recovery (CRh) | Up to 42 months
  Percentage of participants with CRh will be reported based on ELN 2017 response criteria assessment.
Percentage of Participants with CR with Incomplete Recovery (CRi) | Up to 42 months
  Percentage of participants with CRi will be reported based on ELN 2017 response criteria assessment.
Percentage of Participants with CR plus CRh | Up to 42 months
  Percentage of participants with CR plus CRh will be reported based on ELN 2017 response criteria assessment.
Overall Response Rate (ORR) | Up to 42 months
  ORR is defined as percentage of participants with CR, CRh and CRi based on ELN 2017 response criteria assessment.
Percentage of Participants with CR without MRD | Up to 42 months
  Percentage of participants with CR without minimal residual disease (MRD) will be reported and is defined as less than (<) 1 blast or leukemic stem cell in 1,000 leukocytes (MRD level <10^-3).
Percentage of Participants with Negative MRD who Achieved CR, CRh, CRi, or Morphologic Leukemia-free State (MLFS) | Up to 42 months
  Percentage of participants with negative MRD who achieved CR, CRh, CRi, or MLFS will be reported and is defined as < 1 blast or leukemic stem cell in 1,000 leukocytes (MRD level <10^-3).
Cohort 2 and 3: Time to Response | Up to 42 months
  Time to response is defined as time from first dose to achieving the first response of CR, CRh, or CRi.
Cohort 2 and 3: Duration of Response | Up to 42 months
  Duration of response is defined as time from achieving the first response of CR, CRh, or CRi to hematologic relapse or death of any cause.
Cohort 2 and 3: Red Blood Cell (RBC) or Platelet Transfusion Independence | Up to 42 months
  Transfusion independence (RBC or platelets) is defined as a period of greater than or equal to (>=) 56 consecutive days with no transfusion between first dose of study drug and the last dose of study drug +30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Smith, MD, Study Director — OncoVerity, Inc.
Locations (23):
- United States (11):
  - City of Hope, Duarte, California
  - Norton Cancer Institute, Louisville, Kentucky
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Vermont, Burlington, Vermont
  - Wisconsin Medical Center, Milwaukee, Wisconsin
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Toronto, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Germany (3):
  - Universitaetsklinik Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Universitaet Muenchen, München
- Poland (3):
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Instytut Hematologii i Transfuzjologii, Warsaw
- Switzerland (2):
  - INSELSPITAL, Universitätsspital Bern, Bern
  - Kantonsspital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Pabst T, Papayannidis C, Demirkan F, Doronin V, Fogliatto LM, Guttke C, Gyan E, Hamad N, Herrera P, Hultberg A, Jacobs J, Johnson AJ, Langlois A, Ma X, Martinelli G, Arnan M, Muller R, Nottage K, Ofran Y, Ozcan M, Samoilova O, Tolbert JA, Trudel GC, Xiu L, Vey N, Wei AH. Cusatuzumab plus azacitidine in newly diagnosed acute myeloid leukaemia ineligible for intensive chemotherapy (CULMINATE): part one of a randomised, phase 2, dose optimisation study. Lancet Haematol. 2023 Nov;10(11):e902-e912. doi: 10.1016/S2352-3026(23)00207-7. PMID 37914483
- [Derived] Dewulf J, Flieswasser T, Delahaye T, Vangestel C, Miranda A, de Haard H, Jacobs J, Smits E, Van den Wyngaert T, Elvas F. Site-specific 68Ga-labeled nanobody for PET imaging of CD70 expression in preclinical tumor models. EJNMMI Radiopharm Chem. 2023 Apr 24;8(1):8. doi: 10.1186/s41181-023-00194-3. PMID 37093350